CLINICAL TRIAL: NCT03646643
Title: Prospective Elimination Of Distal Coronary Sinus-Left Atrial Connections for Atrial Fibrillation Ablation Trial
Acronym: PRECAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Dr. Saman Nazarian, Associate Professor of Medicine, Cardiac Electrophysiology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 829990
Record Dates: First submitted 2018-08-06; First posted 2018-08-24 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation; Arrhythmias, Cardiac
Keywords: Atrial fibrillation; Coronary sinus-left atrium connection; Ablation
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: The PRECAF study is designed as a randomized, single-blind, small scale pilot study. Enrolled subjects who satisfy all eligibility criteria will then undergo the ablation procedure. Study randomization will be performed in a 1:1 fashion using the Urn Randomization program (https://health.uconn.edu/community-medicine/programs/health-services-research-unit/project-match/urn-randomization/) while balancing sex and AF type (paroxysmal and non-paroxysmal). The master list of study assignments will be kept by the study coordinator in a password protected and encrypted computer. After the ablation procedure, participants will remain in the study for 6 months. A 30-day event monitor will be used for the first month after ablation. Then, regular clinic visits at 6 weeks and 6 months will be arranged after ablation with 12 lead electrocardiogram check-up. In the last month, a 30-day event monitor will again be utilized to detect atrial arrhythmia recurrence.
Who Masked: Participant, Outcomes Assessor
Masking Description: Once patients are enrolled in the study, they will be randomized to arm A: PVI + triggers ablation, or arm B: PVI + triggers ablation + coronary sinus-left atrium connection ablation. Patients will be blinded to the randomization scheme.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVI, non-PV triggers (Active Comparator): Interventions: Atrial fibrillation ablation, including conventional pulmonary vein isolation (PVI) and non-PV triggers ablation.
  Interventions: Procedure: Standard Atrial fibrillation ablation
- PVI, non-PV triggers & CS-LA connection (Active Comparator): Interventions: Atrial fibrillation ablation, including conventional pulmonary vein isolation (PVI) and non-PV triggers ablation in addition to coronary sinus-left atrium connection elimination. Distal coronary sinus pacing will be utilized to localize the earliest connection (aside from septal) from the coronary sinus to the left atrial musculature. Once localized, focal radiofrequency lesions will be applied at the discretion of the investigator until distal coronary sinus to left atrial connections are eliminated.
  Interventions: Procedure: Standard Atrial fibrillation ablation; Procedure: Coronary sinus to left atrium connection elimination

INTERVENTIONS:
Procedure: Standard Atrial fibrillation ablation — The AF ablation procedures should follow the sequence below: Diagnostic catheter placement Electrophysiology study; Transseptal puncture; Left atrial electro-anatomical mapping is required prior to an ablation procedure. Post ablation pacing procedure(s) and/or infusion of cardiac medications to localize triggers/ assess and localize pulmonary vein reconnections (e.g., Adenosine, Isoproterenol 2-20 mcg/min). Study procedure requirements are outlined below: Isolation of all pulmonary veins and Non-pulmonary vein trigger ablation for all patients. Linear ablation lines are only required to treat documented macro-reentry atrial tachycardias and limited to the following targets only: LA roof line, mitral valve isthmus line, LA floor line, right atrial carvotricuspid isthmus linear ablation.
  Other Names: Pulmonary vein isolation; Non-PV triggers ablation
Procedure: Coronary sinus to left atrium connection elimination — Distal coronary sinus pacing will be utilized to localize distal connections between the main coronary sinus body and the left atrium. Focal lesions will be applied to early left atrial activation sites, until no distal coronary sinus to left atrial connections are electrically manifest. If vein of marshall connections to the left atrium are present, differential pacing will be utilized to prove the lack of distal coronary sinus to left atrium connections.
  Arms: PVI, non-PV triggers & CS-LA connection

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmia affecting millions of people in the US and around the world. Over the last 20 years, catheter based AF ablation has been widely adopted offering improved symptom control for many patients worldwide. However, long-term success rates remain suboptimal. Prior work indicates that distal connections between coronary sinus musculature and the left atrium exist and provide a substrate for single or multiple reentry beats as a trigger for atrial fibrillation. In this trial, the investigators will examine the efficacy of elimination of distal connection(s) between coronary sinus and left atrial musculature for suppression of recurrent atrial arrhythmias.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac arrhythmia affecting millions of people in the US and around the world. Over the last 20 years, catheter based AF ablation has been widely adopted. However, long-term success rates fhave been reported to be as low as 50% and 20% for paroxysmal and persistent AF, respectively. To achieve permanent arrhythmia suppression, repeated ablation procedures are often needed. Prior work indicates that distal connections between coronary sinus musculature and the left atrium provide a substrate for single or multiple reentry beats as a trigger for atrial fibrillation. In this prospective randomized trial the investigators will define the efficacy of elimination of distal connections between coronary sinus and left atrial musculature for suppression of recurrent atrial arrhythmias. Patients will be randomly assigned to standard of care ablation (pulmonary vein isolation and non pulmonary vein trigger ablations) alone, or standard of care ablation augmented by distal coronary sinus to left atrial connection elimination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal or persistent atrial fibrillation; AND Undergoing first AF ablation; AND Age ≥ 18 years.

Exclusion Criteria:

* Previous left atrial ablation; Women currently pregnant; Mental or physical inability to take part in the study; Known terminally ill patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-08-18 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2021-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saman Nazarian, M.D., Ph.D, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Information about study subjects will be kept confidential and managed according to the requirements of the Health Insurance Portability and Accountability Act of 1996 (HIPAA). Those regulations require a signed subject authorization informing the subject of the following:
  * What protected health information (PHI) will be collected from subjects in this study
  * Who will have access to that information and why
  * Who will use or disclose that information
  * The rights of a research subject to revoke their authorization for use of their PHI.
  In the event that a subject revokes authorization to collect or use PHI, the investigator, by regulation, retains the ability to use all information collected prior to the revocation of subject authorization. For subjects that have revoked authorization to collect or use PHI, attempts should be made to obtain permission to collect at least vital status (i.e. that the subject is alive) at the end of their scheduled study period.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Recruitment will end when 100 participants are enrolled at Penn. Enrolled subjects who satisfy all eligibility criteria will then undergo the ablation procedure. After the study ablation procedure, participants will be part of the study for 6 months after ablation. A 30-day event monitor will be used for the first month after ablation. Then, regular clinic visits at 6 weeks and 6 months will arranged after ablation with 12 lead electrocardiogram check-up. In the last month, a 30- day event monitor will be set to detect the recurrence of atrial arrhythmias. All data are available and stored for 7 years after the end of the study.

REFERENCES:
- [Result] Kim MH, Lin J, Kreilick C, Foltz Boklage SH. Total costs and atrial fibrillation ablation success or failure in Medicare-aged patients in the United States. Adv Ther. 2010 Sep;27(9):600-12. doi: 10.1007/s12325-010-0060-3. Epub 2010 Aug 9. PMID 20700678
- [Result] Chauvin M, Shah DC, Haissaguerre M, Marcellin L, Brechenmacher C. The anatomic basis of connections between the coronary sinus musculature and the left atrium in humans. Circulation. 2000 Feb 15;101(6):647-52. doi: 10.1161/01.cir.101.6.647. PMID 10673257
- [Result] Huang D, Marine JE, Li JB, Zghaib T, Ipek EG, Sinha S, Spragg DD, Ashikaga H, Berger RD, Calkins H, Nazarian S. Association of Rate-Dependent Conduction Block Between Eccentric Coronary Sinus to Left Atrial Connections With Inducible Atrial Fibrillation and Flutter. Circ Arrhythm Electrophysiol. 2017 Jan;10(1):e004637. doi: 10.1161/CIRCEP.116.004637. PMID 28039281
- [Result] Antz M, Otomo K, Arruda M, Scherlag BJ, Pitha J, Tondo C, Lazzara R, Jackman WM. Electrical conduction between the right atrium and the left atrium via the musculature of the coronary sinus. Circulation. 1998 Oct 27;98(17):1790-5. doi: 10.1161/01.cir.98.17.1790. PMID 9788835
- [Derived] Kuo L, Frankel DS, Lin A, Arkles J, Hyman M, Santangeli P, Marchlinski FE, Nazarian S. PRECAF Randomized Controlled Trial. Circ Arrhythm Electrophysiol. 2021 Jan;14(1):e008993. doi: 10.1161/CIRCEP.120.008993. Epub 2020 Dec 10. PMID 33301361

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study is a single-center, randomized, controlled trial, enrolling drug-refractory symptomatic patients who presented for first-time atrial fibrillatoin ablation at the Hospital of the University of Pennsylvania between August 2018 and August 2019 (PRECAF [Prospective Elimination of Distal Coronary Sinus to Left Atrial Connection for Atrial Fibrillation Ablation])
Groups:
- PVI, Non-PV Triggers Ablation: Interventions: Atrial fibrillation ablation, including conventional pulmonary vein isolation (PVI) and non-PV triggers ablation.
  Standard Atrial fibrillation ablation: The AF ablation procedures should follow the sequence below: Diagnostic catheter placement Electrophysiology study; Transseptal puncture; Left atrial electro-anatomical mapping is required prior to an ablation procedure. Post ablation pacing procedure(s) and/or infusion of cardiac medications to localize triggers/ assess and localize pulmonary vein reconnections (e.g., Adenosine, Isoproterenol 2-20 mcg/min). Study procedure requirements are outlined below: Isolation of all pulmonary veins and Non-pulmonary vein trigger ablation for all patients. Linear ablation lines are only required to treat documented macro-reentry atrial tachycardias and limited to the following targets only: LA roof line, mitral valve isthmus line, LA floor line, right atrial carvotricuspid isthmus linear ablation.
- PVI, Non-PV Triggers Ablation & Elimination of Distal CS-LA Connection: Interventions: AF ablation, including conventional PVI and non-PV triggers ablation in addition to coronary sinus (CS)-left atrium (LA) connection elimination. Distal CS pacing will be utilized to localize the earliest connection (aside from septal) from the CS to the LA musculature. Once localized, focal radiofrequency lesions will be applied at the discretion of the investigator until distal CS to LA connections are eliminated.
  If vein of Marshall connections to the LA are present, differential pacing will be utilized to prove the lack of distal CS to LA connections.
  Post ablation pacing procedure(s) and/or infusion of cardiac medications to localize triggers/ assess and localize pulmonary vein reconnections (e.g., Adenosine, Isoproterenol 2-20 mcg/min) Linear ablation lines are only required to treat documented macro-reentry atrial tachycardias and limited to the following targets only: LA roof line, mitral valve isthmus line, LA floor line, right atrial carvotricuspid isthmus linear ablation.
Period: Overall Study
Arm/Group | PVI, Non-PV Triggers Ablation | PVI, Non-PV Triggers Ablation & Elimination of Distal CS-LA Connection
Started | 17 | 18
Completed | 15 | 15
Not Completed | 2 | 3
Not completed — Not yet achieved 6 months study follow-up at the time of analysis | 2 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: The study is a single-center, randomized, controlled trial, enrolling drug-refractory symptomatic patients who presented for first-time AF ablation at the Hospital of the University of Pennsylvania between August 2018 and August 2019.
Groups:
- PVI, Non-PV Triggers & CS-LA Connection: Interventions: Atrial fibrillation ablation, including conventional pulmonary vein isolation (PVI) and non-PV triggers ablation in addition to coronary sinus-left atrium connection elimination.
  Isolation of all pulmonary veins and non-pulmonary vein trigger ablation for all patients. Linear ablation lines are only required to treat documented macro-reentry atrial tachycardias and limited to the following targets only: LA roof line, mitral valve isthmus line, LA floor line, right atrial carvotricuspid isthmus linear ablation.
  In persistent atrial fibrillation patients, cardioversion can be performed if rhythm cannot be restored to sinus rhythm after PVI with/without posterior wall box isolation. Then, distal coronary sinus pacing will be utilized to localize the earliest connection (aside from septal) from the coronary sinus to the left atrial musculature. Once localized, focal radiofrequency lesions will be applied at the discretion of the investigator until distal coronary sinus to left atrial connections are eliminated. If vein of marshall connections to the left atrium are present, differential pacing will be utilized to prove the lack of distal coronary sinus to left atrium connections.
- Total: Total of all reporting groups
Arm/Group | PVI, Non-PV Triggers | PVI, Non-PV Triggers & CS-LA Connection | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Categorical [Count of Participants; unit: Participants] — Population: The study is a single-center, randomized, controlled trial, enrolling drug-refractory symptomatic patients who presented for first-time ablation at the Hospital of the University of Pennsylvania between August 2018 and August 2019. Atrial arrhythmia recurrence at follow-up was reported with a time-to-event analysis with censoring on November 20, 2019.
  Participants
    number analyzed (Participants) | 15 | 15 | 30
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 5 | 8 | 13
    >=65 years | 10 | 7 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The study is a single-center, randomized, controlled trial, enrolling drug-refractory symptomatic patients who presented for first-time ablation at the Hospital of the University of Pennsylvania between August 2018 and August 2019. Atrial arrhythmia recurrence at follow-up was reported with a time-to-event analysis with censoring on November 20, 2019.
  years
    number analyzed (Participants) | 15 | 15 | 30
    (all) | 66.7 (6.1) | 64.6 (8.3) | 65.6 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The study is a single-center, randomized, controlled trial, enrolling drug-refractory symptomatic patients who presented for first-time ablation at the Hospital of the University of Pennsylvania between August 2018 and August 2019. Atrial arrhythmia recurrence at follow-up was reported with a time-to-event analysis with censoring on November 20, 2019. Four patients had not achieve 6 months study follow-up at the time of analysis; there was one patient loss follow-up.
  Participants
    number analyzed (Participants) | 15 | 15 | 30
    Female | 9 | 5 | 14
    Male | 6 | 10 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The study is a single-center, randomized, controlled trial, enrolling drug-refractory symptomatic patients who presented for first-time ablation at the Hospital of the University of Pennsylvania between August 2018 and August 2019. Atrial arrhythmia recurrence at follow-up was reported with a time-to-event analysis with censoring on November 20, 2019. Four patients had not achieve 6 months study follow-up at the time of analysis; there was one patient loss follow-up.
  Participants
    number analyzed (Participants) | 15 | 15 | 30
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 1 | 2
    White | 13 | 13 | 26
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: The study is a single-center, randomized, controlled trial, enrolling drug-refractory symptomatic patients who presented for first-time ablation at the Hospital of the University of Pennsylvania between August 2018 and August 2019. Atrial arrhythmia recurrence at follow-up was reported with a time-to-event analysis with censoring on November 20, 2019. Four patients had not achieve 6 months study follow-up at the time of analysis; there was one patient loss follow-up.
  Participants
    United States: number analyzed (Participants) | 15 | 15 | 30
    United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Recurrence Rate of Atrial Arrhythmias
Description: The primary endpoint of the study is recurrence rate of atrial arrhythmia following ablation. The primary endpoint will be assessed using survival statistical models measuring time to failure among the two study arms. Failure is defined as a non-self-terminating bout of atrial fibrillation, atrial flutter, or atrial tachycardia >30 seconds in duration following the 90-day post-ablation blanking period. If no AF occurs during the study period, censoring will occur at 180±45 days post-ablation.
Time Frame: Time to atrial arrhythmia recurrence will be recorded as time to the first ECG or monitor that shows atrial arrhythmia recurrence between the end of the blanking period (90 days post ablation) and the end of the study (180±45 days post ablation).
Measure: Number; unit: participants
Groups:
- PVI, Non-PV Triggers Ablation Isolation and Non-pulmonary Vein Trigger Ablation: Interventions: Atrial fibrillation ablation, including conventional pulmonary vein isolation (PVI) and non-PV triggers ablation.
  Standard Atrial fibrillation ablation: The AF ablation procedures should follow the sequence below: Diagnostic catheter placement Electrophysiology study; Trans-septal puncture; Left atrial electro-anatomical mapping is required prior to an ablation procedure. Post ablation pacing procedure(s) and/or infusion of cardiac medications to localize triggers/ assess and localize pulmonary vein reconnections (e.g., Adenosine, Isoproterenol 2-20 mcg/min). Study procedure requirements are outlined below: Isolation of all pulmonary veins and Non-pulmonary vein trigger ablation for all patients. Linear ablation lines are only required to treat documented macro-reentry atrial tachycardias and limited to the following targets only: LA roof line, mitral valve isthmus line, LA floor line, right atrial carvotricuspid isthmus linear ablation.
- PVI, Non-PV Triggers Ablation+Elimination of Distal CS to LA Connections: Interventions: AF ablation, including conventional PVI and non-PV triggers ablation in addition to coronary sinus (CS)-left atrium (LA) connection elimination. Distal CS pacing will be utilized to localize the earliest connection (aside from septal) from the CS to the LA musculature. Once localized, focal radiofrequency lesions will be applied at the discretion of the investigator until distal CS to LA connections are eliminated. If vein of Marshall connections to the LA are present, differential pacing will be utilized to prove the lack of distal CS to LA connections.
  If persistent atrial fibrillation cannot be restored to sinus rhythm after PVI, cardioversion with/without posterior wall box isolation can be performed. Then, non-PV triggers can be evaluated and distal CS-pacing can be ultilized to identify the CS to LA connection.
  Post ablation pacing procedure(s) and/or infusion of cardiac medications to localize triggers/ assess and localize pulmonary vein reconnections (e.g., Adenosine, Isoproterenol 2-20 mcg/min).
  Linear ablation lines are only required to treat documented macro-reentry atrial tachycardias and limited to the following targets only: LA roof line, mitral valve isthmus line, LA floor line, right atrial carvotricuspid isthmus linear ablation.
Arm/Group | PVI, Non-PV Triggers Ablation Isolation and Non-pulmonary Vein Trigger Ablation | PVI, Non-PV Triggers Ablation+Elimination of Distal CS to LA Connections
Number analyzed (Participants) | 15 | 15
participants
  No Atrial Arrhythmia Recurrence | 8 | 14
  Atrial Arrhythmia Recurrence | 7 | 1
Statistical Analysis 1: Comparison: PVI, Non-PV Triggers Ablation Isolation and Non-pulmonary Vein Trigger Ablation vs PVI, Non-PV Triggers Ablation+Elimination of Distal CS to LA Connections; Power calculation: assuming alpha 0.05, power 0.8, 1:1 randomization, and estimated relative risk of 14.4 for AF susceptibility with rate-dependent CS-LA conduction block, we anticipated a minimum sample size of 6 patients per group would be necessary to detect a difference using the log-rank test. Additional patients were recruited to account for potential losses to follow-up and a smaller detectable difference; Test type: Superiority; p = 0.047, Log Rank — A priori threshold <0.05. Multiple comparisons adjustments: not needed; Hazard Ratio (HR) = 0.12, 95% CI 2-sided [0.02 to 0.97] — The distal CS to LA connection elimination group had fewer recurrences (6.7%) compared with the standard group (46.7%), which translated to an 88% lower hazard of recurrence compared with the standard group

ADVERSE EVENTS:
Time Frame: The study enrolled drug-refractory symptomatic AF patients who presented for first-time ablation at the Hospital of the University of Pennsylvania between August 2018 and August 2019. Atrial arrhythmia recurrence at follow-up was reported with a time-to-event analysis with censoring on November 20, 2019. Regular clinic visits at 6 weeks and 6 months post-ablation were arranged and adverse events were recorded.
Description: One patient was readmitted with pericarditis. Pericardiocentesis was performed with drainage of 200 mL serous pericardial effusion 16 days following ablation, which included PV isolation (35 minutes radiofrequency [RF] time), mitral isthmus line (10 minutes RF time), and distal CS to LA connection elimination (1.5 minutes RF time)--no clearly attributed to the strategy of distal CS to LA connection elimination. The patient recovered and was discharged on anticoagulation without further sequela.
Groups:
- PVI, Non-PV Triggers & CS-LA Connection: Interventions: AF ablation, including conventional PVI and non-PV triggers ablation in addition to coronary sinus (CS)-left atrium (LA) connection elimination. Distal CS pacing will be utilized to localize the earliest connection (aside from septal) from the CS to the LA musculature. Once localized, focal radiofrequency lesions will be applied at the discretion of the investigator until distal CS to LA connections are eliminated.
  If vein of Marshall connections to the LA are present, differential pacing will be utilized to prove the lack of distal CS to LA connections.
  Post ablation pacing procedure(s) and/or infusion of cardiac medications to localize triggers/ assess and localize pulmonary vein reconnections (e.g., Adenosine, Isoproterenol 2-20 mcg/min) Linear ablation lines are only required to treat documented macro-reentry atrial tachycardias and limited to the following targets only: LA roof line, mitral valve isthmus line, LA floor line, right atrial carvotricuspid isthmus linear ablation.
Arm/Group | PVI, Non-PV Triggers | PVI, Non-PV Triggers & CS-LA Connection
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PVI, Non-PV Triggers (N=15) | PVI, Non-PV Triggers & CS-LA Connection (N=15)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) — One patient presented with pericarditis requiring pericardiocentesis of 200 mL serous effusion 16 days after PV, mitral annular and CS to LA connection ablation. The patient was discharged on anticoagulation and without further sequela.

LIMITATIONS AND CAVEATS:
(1) A single-center pilot study with a relatively small sample size; (2) 40% of patients underwent insertable cardiac monitor implantation; (3) Of patients without insertable monitors, 56% had 30-days wearable monitor pre-ablation, during the 1st & 6th-month after ablation. (4) 44% had follow-up for detection of atrial arrhythmia recurrences based upon symptom or pulse check prompted monitors and ECGs during clinic visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/43/NCT03646643/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/43/NCT03646643/ICF_001.pdf